CLINICAL TRIAL: NCT05656066
Title: The Effects of Vibration and Pressure Interventions on Pain, Fear and Anxiety in Pediatric Patients Coming to the Emergency Department for Intramuscular Injection
Brief Title: The Effects of Vibration and Pressure Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ıntramuscular
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Anxiety
Keywords: anxiety; fear; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, and experimental design
Who Masked: Participant
Masking Description: Participants will not know which group in. Researcher and nurse will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Vibration Intervention Group (VI) (Experimental): After the injection area was determined in the VI group, the vibration device was held for 30 seconds in the area to be injected, then the injection was applied by pulling up 3 cm while the device was operating.
  Interventions: Behavioral: The Vibration Intervention
- The Pressure Intervention Group (Experimental): After the injection area was determined in the PI group, 30 seconds light pressure was applied with the thumb and then the injection was given
  Interventions: Behavioral: The Pressure Intervention
- The Control Group (No Intervention): The routine IM injection was applied to the children in the control group.

INTERVENTIONS:
Behavioral: The Vibration Intervention — The vibration frequency of the massager, which accelerates blood circulation, is 6000 / min, it works with a 1.5 volt battery. Can be used easily with one hand. The vibration simulator design is based on the gate-control theory, which allows for a reduction in the perceived amount of pain experienced during injection by closing the pain gate in the spinal cord in creating a stimulus on the skin.
  Arms: The Vibration Intervention Group (VI)
Behavioral: The Pressure Intervention — Pressure was placed in the ıntramuscular area properly 30 seconds before injection. Then the injection process was completed.
  Arms: The Pressure Intervention Group

SUMMARY:
This study aimed to evaluate two methods (pressure and vibration intervention) used to reduce pain during IM injections in children.

DETAILED DESCRIPTION:
Objectives: This study was conducted to evaluate the effects of the Vibration and Pressure Intervention for reducing pain during intramuscular (IM) injections in children.

Design: The study was conducted via a randomized controlled design. Setting: The study population consisted of children in the five to 10 age group admitted to the emergency department of a public hospital (Samsun Education and Research Hospital) between August 2022 and October 2022 and who received an IM injection as part of the medical treatment in child emergency department.

Interventions: The study data were collected from the children, who were divided into Vibration Intervention group, Pressure Intervention group, and control groups.

Main outcome measures: The children's pre-procedure fear and anxiety levels were evaluated using the Children's Fear Scale (CFS), and Children' Anxiety Meter State. Then, their pain levels during the procedure were evaluated using the Wong-Baker FACES Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* had no diagnosed physical or mental disability or chronic illness;
* had no communication problems;
* received single injection,
* required seftriakson group of antibiotics for standardization; and received vastus lateralis muscle injection during the study.

Exclusion Criteria:

* Parents who were unable to collaborate in the fear and pain evaluation,
* overweight or underweight children (under the third or above the 97th percentile),
* children with any incision or scar tissue in the injection area,
* children who received a sedative, analgesic, or narcotic drugs (based on expert opinion) six hours before the procedure on the basis of parental statements and medical history

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Children's Fear Scale (CFS) | during procedure
  The Children's Fear Scale (CFS) is a scale used to assess the level of anxiety in children. The scale is a visual measurement tool with scores ranging from 0-4 points. It consists of five facial expressions, ranging from a neutral to a frightened expression, and is suitable for use with children aged 5-10 years (Inan & Inal, 2019; McMurtry, Noel, Chambers, & McGrath, 2011; Özalp Gerçeker, Ayar, Özdemir, & Bektaş, 2018). The evaluation of the Turkish psychometric properties of the scale, which was developed by McMurty et al. for paediatric patients, was conducted by Özalp Gerçeker et al. (2018), and the scale was translated into the Turkish language (Özalp Gerçeker et al., 2018). The CFS has demonstrated good evidence of test-retest (r = 0.76, p < 0.001), and inter-rater (0.51, P < 0.001) reliability, as well as construct validity, (rs ¼ when used with children (McMurtry vd., 2011
The Children's Anxiety Meter-State (CAM-S) | during procedure
  The Children's Anxiety Meter-State (CAM-S) assesses children's anxiety at medical procedures. It is drawn like a thermometer with a bulb at the bottom. It includes horizontal lines going up to the top (0-10). Children are asked to mark their feelings "right now" to measure state anxiety (Kleiber & Mccarthy, 2006). CAM-S was validated in children aged 4-10 years during an intravenous procedure. It is significantly associated with all parent measures and observed distress ratings (Ersig et al., 2013). Gerçeker et al. (2018) conducted the psychometric properties of CAM-S in the Turkish population. They revealed a significant negative correlation between the CAM-S scores and children's ages (β = 0.340, p < .001).
Wong-Baker FACES Rating Scale | during procedure
  It is a horizontal scale developed by Wong and Baker in 1983 for children over 3 years of age who can express themselves. In this scale, pain scores are given to faces according to numerical values. The lowest score is "0" and the highest score is "10". As the score obtained from the scale increases, the severity of pain increases. During the application of the scale, it is stated to the child that each of the facial expressions belongs to a person. It is stated that the child who has no pain expresses a happy face, while the child who has a little or a lot of pain during the procedure has sad faces.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatice Uzşen, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drago LA, Singh SB, Douglass-Bright A, Yiadom MY, Baumann BM. Efficacy of ShotBlocker in reducing pediatric pain associated with intramuscular injections. Am J Emerg Med. 2009 Jun;27(5):536-43. doi: 10.1016/j.ajem.2008.04.011. PMID 19497458
- [Background] Bilge S, Aydin A, Gun C, Aldinc H, Acar YA, Yaylaci S, Cinar O, Balci V. Comparison of the efficacy of ShotBlocker and cold spray in reducing intramuscular injection-related pain in adults. A prospective, randomized, controlled trial. Saudi Med J. 2019 Oct;40(10):996-1002. doi: 10.15537/smj.2019.10.24322. PMID 31588477